CLINICAL TRIAL: NCT05237284
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of SAR443820 in Adult Participants With Amyotrophic Lateral Sclerosis, Followed by an Open-label Extension
Brief Title: Phase 2 Study for SAR443820 in Participants With Amyotrophic Lateral Sclerosis (ALS)
Acronym: HIMALAYA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated as its Part A did not meet the primary endpoint.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT16970; U1111-1263-5766 (Registry Identifier: ICTRP); 2023-509442-36-00 (Registry Identifier: CTIS); 2021-004156-42 (EudraCT Number)
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAR443820 (Experimental): twice daily (BID) oral SAR443820
  Interventions: Drug: SAR443820
- Placebo (Placebo Comparator): twice daily (BID) oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR443820 — Tablet oral
  Arms: SAR443820
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
This was a parallel treatment, Phase 2, randomized, double-blind study to assess the efficacy, safety, tolerability, PK, and PD of twice daily (BID) oral SAR443820 compared with placebo in male and female participants, 18 to 80 years of age with ALS followed by an open-label, long-term extension period.

Study ACT16970 consisted of 2 parts (A and B) as follows:

Part A was a 24-week, double blind, placebo-controlled part, preceded by a screening period of up to 4 weeks before Day 1.

On Day 1 of Part A, participants were randomized in a 2:1 ratio to the SAR443820 treatment arm or matching placebo arm as listed below:

* Treatment arm: SAR443820, BID
* Placebo arm: Placebo, BID

Randomization was stratified by the geographic region of the study site, region of ALS onset (bulbar vs other areas), use of riluzole (yes vs no), use of edaravone (yes vs no) and use of the combination of sodium phenylbutyrate and taurursodiol (named Relyvrio in the United States of America [USA] and Albrioza in Canada) (yes vs no). Participants attended in-clinic study assessments at baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 16, Week 20, Week 21, Week 22, Week 23, and Week 24. All ongoing participants at Week 24 rolled to open-label extension Part B. The Week 24 Visit was the end of Part A and the beginning of Part B.

Part B was an open-label, long-term extension period that starts from Week 24 and continues up to Week 106. The objectives of Part B were to provide extended access to SAR443820 participants in Part A and to further evaluate the safety and efficacy of long-term SAR443820 treatment. The treatment assignment of participants at randomization in Part A remained blinded to Investigators, participants, and site personnel until the end of Part B. Every participant, except those who discontinued Investigational Medicinal Product (IMP) treatment permanently in Part A, received BID oral tablets of SAR443820 in Part B.

DETAILED DESCRIPTION:
The study duration included an up to 4-week screening period, 24-week double-blind treatment period in Part A, 80-week open-label treatment period in Part B and 2-week post-treatment follow-up period, with a maximum total study duration of 110 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, clinically probable ALS, clinically probable laboratory supported ALS, or clinically definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria
* Time since onset of first symptom of ALS ≤2 years.
* Slow Vital Capacity (SVC) ≥60% of the predicted value.
* Had to be able to swallow the study tablets at the screening visit.
* Either not currently receiving riluzole or on a stable dose of riluzole for at least 4 weeks before the screening visit. Participants receiving riluzole were expected to remain on the same dose throughout the duration of the study.
* Either not currently receiving edaravone or on the approved standard schedule of edaravone treatment. Participants receiving edaravone had to have completed at least 1 cycle of treatment before the screening visit and were expected to continue edaravone treatment throughout the duration of the study.
* Either not currently receiving the combination of sodium phenylbutyrate and taurursodiol or on the approved standard schedule of the combination of sodium phenylbutyrate and taurursodiol treatment for at least 4 weeks before the screening visit. Participants receiving the combination of sodium phenylbutyrate and taurursodiol were expected to remain on the approved standard schedule throughout the duration of the study.
* Participants with a body weight no less than 45 kg and body mass index no less than 18 kg/m2 at the screening visit
* Female participants with childbearing potential were eligible to participate if they were not pregnant or breastfeeding and agreed to use adequate contraceptive method during study intervention period and for at least 32 days after the last dose of study drug.
* Male participants had to agree to use highly effective contraceptive method during the study period and for at least 92 days following their last dose of the study drug. Male participants were not donate sperms for the duration of study and 92 days after last dose of study drug.

Exclusion Criteria:

* A history of seizure (History of febrile seizure during childhood was allowed).
* Having central IV lines, such as a peripherally inserted central catheter (PICC XE ' PICC ' \f Abbreviation \t 'peripherally inserted central catheter' ) or midline or portacath lines.
* With significant cognitive impairment, psychiatric disease, other neurodegenerative disorder (eg, Parkinson disease or AD), substance abuse other causes of neuromuscular weakness, or any other condition that would make the participants unsuitable for participating in the study or could interfere with assessment or completing the study in the opinion of the Investigator.
* History of recent serious infection (eg, pneumonia, septicemia) within 4 weeks of the screening visit; infection requiring hospitalization or treatment with IV antibiotics, antivirals, or antifungals within 4 weeks of screening; or chronic bacterial infection (such as tuberculosis) deemed unacceptable as per the Investigator's judgment.
* With active herpes zoster infection within 2 months prior to the screening visit.
* A documented history of attempted suicide within 6 months prior to the screening visit, present with suicidal ideation of category 4 or 5 on the Columbia Suicide Severity Rating Scale (CSSRS) , or in the Investigator's judgment are at risk for a suicide attempt.
* History of unstable or severe cardiac, pulmonary, oncological, hepatic, or renal disease or another medically significant illness other than ALS precluding their safe participation in this study.
* Participants who were pregnant or were currently breastfeeding.
* A known history of allergy to any ingredients of SAR443820.
* Currently or previously treated with any strong or moderate CYP3A4 inhibitors or strong CYP3A4 inducers within the specified washout period before the screening visit.
* Received a live vaccine within 14 days before the screening visit.
* Participants with concurrent participation in any other interventional clinical study or who had received treatment with another investigational drug (eg sodium phenylbutyrate or taurursodiol ) within 4 weeks or 5 halflives of the investigational agent before the screening visit, whichever is longer.
* Participants who had received stem cell or gene therapy for ALS at any time in the past.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3.0 × upper limit of normal (ULN)
* Bilirubin >1.5 × ULN unless the participant had documented Gilbert syndrome (isolated bilirubin >1.5 × ULN was acceptable if bilirubin was fractionated and direct bilirubin is <35%)
* Serum albumin <3.5 g/dL
* Estimated glomerular filtration rate <60 mL/min/1.73 m2 (Modification of Diet in Renal Disease [MDRD])

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (63):
- United States (17):
  - UC San Diego Health Site Number : 8400022, La Jolla, California
  - USC Site Number : 8400008, Los Angeles, California
  - University of California Irvine Site Number : 8400012, Orange, California
  - California Pacific Medical Center Site Number : 8400015, San Francisco, California
  - University of Colorado Site Number : 8400025, Aurora, Colorado
  - Georgetown University Medical Center Site Number : 8400020, Washington D.C., District of Columbia
  - Mayo Clinic Site Number : 8400029, Jacksonville, Florida
  - AdventHealth Medical Group - Neurology at Winter Park Site Number : 8400006, Winter Park, Florida
  - Northwestern Medical Group, Department of Neurology Site Number : 8400003, Chicago, Illinois
  - Johns Hopkins University Site Number : 8400028, Baltimore, Maryland
  - Massachusetts General Hospital Site Number : 8400001, Boston, Massachusetts
  - Mount Sinai - Union Square Site Number : 8400002, New York, New York
  - Penn State Milton S. Hershey Medical Center Site Number : 8400004, Hershey, Pennsylvania
  - University of Pennsylvania Site Number : 8400021, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital Site Number : 8400014, Philadelphia, Pennsylvania
  - University of Utah Site Number : 8400009, Salt Lake City, Utah
  - Froedtert Hospital & Medical College of Wisconsin Site Number : 8400010, Milwaukee, Wisconsin
- Investigational Site Number : 0560001, Leuven, Belgium
- Canada (6):
  - Investigational Site Number : 1240004, Edmonton, Alberta
  - Investigational Site Number : 1240007, Hamilton, Ontario
  - Investigational Site Number : 1240006, London, Ontario
  - Investigational Site Number : 1240008, Toronto, Ontario
  - Investigational Site Number : 1240002, Montreal, Quebec
  - Investigational Site Number : 1240001, Québec
- China (6):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560003, Chengdu
  - Investigational Site Number : 1560005, Guangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560004, Wuhan
  - Investigational Site Number : 1560006, Xi'an
- France (6):
  - Investigational Site Number : 2500007, Caen
  - Investigational Site Number : 2500006, Lille
  - Investigational Site Number : 2500002, Marseille
  - Investigational Site Number : 2500003, Montpellier
  - Investigational Site Number : 2500004, Tours
  - Investigational Site Number : 2500005, Vandœuvre-lès-Nancy
- Germany (7):
  - Investigational Site Number : 2760004, Berlin
  - Investigational Site Number : 2760003, Dresden
  - Investigational Site Number : 2760008, Haag in OB
  - Investigational Site Number : 2760005, Hanover
  - Investigational Site Number : 2760002, Lübeck
  - Investigational Site Number : 2760001, Ulm
  - Investigational Site Number : 2760009, Würzburg
- Italy (3):
  - Investigational Site Number : 3800001, Milan
  - Investigational Site Number : 3800004, Milan
  - Investigational Site Number : 3800002, Torino
- Japan (6):
  - Investigational Site Number : 3920003, Nagoya, Aichi-ken
  - Investigational Site Number : 3920004, Ichikawa-shi, Chiba
  - Investigational Site Number : 3920006, Tokushima, Tokushima
  - Investigational Site Number : 3920005, Fuchu-shi, Tokyo
  - Investigational Site Number : 3920001, Ōta-ku, Tokyo
  - Investigational Site Number : 3920002, Koshi-shi
- Investigational Site Number : 5280001, Utrecht, Netherlands
- Poland (2):
  - Investigational Site Number : 6160001, Krakow
  - Investigational Site Number : 6160002, Ksawerów
- Spain (4):
  - Investigational Site Number : 7240005, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240001, Valencia
- Sweden (2):
  - Investigational Site Number : 7520002, Stockholm
  - Investigational Site Number : 7520001, Umeå
- United Kingdom (2):
  - Investigational Site Number : 8260002, Plymouth, Devon
  - Investigational Site Number : 8260003, Stoke-on-Trent, Staffordshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Hincelin-Mery A, Nicolas X, Cantalloube C, Pomponio R, Lewanczyk P, Benamor M, Ofengeim D, Krupka E, Hsiao-Nakamoto J, Eastenson A, Atassi N. Safety, pharmacokinetics, and target engagement of a brain penetrant RIPK1 inhibitor, SAR443820 (DNL788), in healthy adult participants. Clin Transl Sci. 2024 Jan;17(1):e13690. doi: 10.1111/cts.13690. Epub 2023 Dec 11. PMID 38010108
- See also: ACT16970 (Himalaya study)-Amyotrophic Lateral Sclerosis website — https://www.sanofistudies.com/ALS

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is double-blind followed by an open-label extension, 2 parts: Part (A and B) conducted at 63 investigational sites in 13 countries. A total of 397 participants were screened between 13 Apr 2022 and 17 July 2023, of which 92 were screen failures. Screen failures were due to not meeting the eligibility criteria.
Pre-assignment Details: The study consisted of a screening period (up to 4 weeks prior to randomization), treatment period (a 24-week double-blinded in Part A, an 80-week open-label in Part B), and a 2-week post-treatment follow up period, with a maximum total study duration of 110 weeks. The study was terminated as Part A did not meet the primary endpoint.
Groups:
- Part A: Placebo: Participants received placebo matching to SAR443820 tablet orally twice a day (BID) for 24 weeks in Part A.
- Part A: SAR443820: Participants received SAR443820 20 milligram (mg) tablet orally BID for 24 weeks in Part A.
- Part B: Placebo/SAR443820: Participants who had received placebo matching to SAR443820 tablet in Part A, continued to receive SAR443820 20 mg tablet orally BID for 80 weeks during Part B.
- Part B: SAR443820/SAR443820: Participants who had received SAR443820 tablet in Part A, continued to receive SAR443820 20 mg tablet orally BID for 80 weeks during Part B.
Period: Part A (Double-blind Period: 24 Weeks)
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Started | 102 | 203 | 0 | 0
Randomized and Treated (Participants who had received at least 1 dose of the study treatment.) | 102 | 202 | 0 | 0
Completed | 88 | 167 | 0 | 0
Not Completed | 14 | 36 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 13 | 0 | 0
Not completed — Poor compliance to protocol | 0 | 1 | 0 | 0
Not completed — Adverse Event | 6 | 20 | 0 | 0
Period: Part B (Open-label Period: 80 Weeks)
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Started | 0 | 0 | 88 | 167
Treated (Participants who had received at least 1 dose of the study treatment.) | 0 | 0 | 79 | 136
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 88 | 167
Not completed — Other | 0 | 0 | 0 | 3
Not completed — Study terminated by sponsor | 0 | 0 | 64 | 126
Not completed — Withdrawal by Subject | 0 | 0 | 11 | 21
Not completed — Poor compliance to protocol | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 13 | 16

BASELINE CHARACTERISTICS:
Population: Randomized population=all participants from screened population who had been allocated to a randomized study treatment by interactive response technology (IRT) regardless of whether study treatment was received. Participants from Part A were allowed to transition to Part B per the study design hence baseline characteristics collected at the beginning of the study applies to both Part A and Part B.
Groups:
- Part A: Placebo: Participants received placebo matching to SAR443820 tablet orally BID for 24 weeks in Part A.
- Part A: SAR443820: Participants received SAR443820 20 mg tablet orally BID for 24 weeks in Part A.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: SAR443820 | Total
Number analyzed (Participants) | 102 | 203 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (11.5) | 57.0 (11.6) | 56.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 84 | 122
  Male | 64 | 119 | 183
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 26 | 52 | 78
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 1 | 3 | 4
  White | 69 | 126 | 195
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 21 | 26
Baseline Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) Total Score [Mean (Standard Deviation); unit: score on a scale] — The ALSFRS-R is an instrument to evaluate the functional status of participants with amyotrophic lateral sclerosis (ALS). It consists of 12 items across 4 sub-domains of bodily function: bulbar, fine motor, gross motor, and breathing. Each item was scored on an ordinal scale from 0 (total loss of function) to 4 (no loss of function). The total scores was the sum of the individual items score and it ranges from 0 to 48, with a higher score indicating better function. Baseline was defined as the Day 1 pre-dose value. Population: Only participants with data collected at specified timepoints are reported.
  score on a scale
    number analyzed (Participants) | 100 | 199 | 299
    (all) | 36.23 (5.00) | 35.97 (4.41) | 36.06 (4.61)

OUTCOME MEASURES:

1. Secondary Outcome: Part A: Combined Assessment of the Function and Survival Score at Week 24
Description: The CAFS at Week 24 is a composite endpoint based on time to earlier occurrence of death or permanent assisted ventilation (>22 hours a day for >7 consecutive days) and change from baseline in ALSFRS-R score up to Week 24. ALSFRS-R is a rating scale where 12 functions are rated on 5-point scales (from 0 to 4) with a maximum score of 48 (sum of all 12 items), with a higher score indicating better function. Each participant's outcome was compared to every other participant's outcome by time to death or permanent assisted ventilation and change on ALSFRS-R if survived without permanent assisted ventilation, assigned a score which is sum of comparisons (+1 [better], 0 [tie], -1 [worse]), and summed scores were ranked, from 1 to 296 (mITT population) lowest rank corresponds to participant who died first and highest rank to 1 with best ALSFRS-R outcome among those who survived. A higher rank is considered a better outcome.
Time Frame: Week 24
Population: The mITT population consisted of all randomized participants who either died or had available baseline and at least 1 post-baseline ALSFRS-R assessment. Only participants with data collected at Week 24 is reported. The study was terminated prematurely since the Part A did not meet the primary endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 100 | 196
score on a scale | 151.19 (90.71) | 147.13 (83.06)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: SAR443820; CAFS at Week 24 was analyzed using the Wilcoxon-Mann-Whitney test to compare mean scores between the treatment groups at Week 24; Test type: Superiority; p = 0.6999, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Combined Assessment of the Function and Survival Score at Weeks 76 and 104
Description: The CAFS at Weeks 76 and 106 is a composite endpoint based on time to earlier occurrence of death or permanent assisted ventilation (>22 hours a day for >7 consecutive days) and change from baseline in ALSFRS-R score up to Weeks 76 and 104. ALSFRS-R is a rating scale where 12 functions are rated on 5-point scales (from 0 to 4) with a maximum score of 48 (sum of all 12 items), with a higher score indicating better function. Each participant's outcome was compared to every other participant's outcome by time to death or permanent assisted ventilation and change on ALSFRS-R if survived without permanent assisted ventilation, assigned a score which is sum of comparisons (+1 [better], 0 [tie], -1 [worse]), and summed scores were ranked, from 1 to 296 (mITT population) lowest rank corresponds to participant who died first and highest rank to 1 with best ALSFRS-R outcome among those who survived. A higher rank is considered a better outcome.
Time Frame: Weeks 76 and 104
Population: The mITT population consisted of all randomized participants who either died or had available baseline and at least 1 post-baseline ALSFRS-R assessment. Only participants with data collected at specified timepoints are reported. The study was terminated prematurely since the Part A did not meet the primary endpoint. The data for Week 104 was not collected. All participants who had either early termination or who did not enter Part B, were also included in Week 76 analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo/SAR443820: Participants who had received placebo matching to SAR443820 tablet in Part A for 24 weeks, continued to receive SAR443820 20 mg tablet orally BID for 80 weeks during Part B.
  All death participants were automatically included in this analysis, irrespective whether they reached Week 76 or not.
- SAR443820/SAR443820: Participants who had received SAR443820 tablet in Part A for 24 weeks, continued to receive SAR443820 20 mg tablet orally BID for 80 weeks during Part B.
  All death participants were automatically included in this analysis, irrespective whether they reached Week 76 or not.
Arm/Group | Placebo/SAR443820 | SAR443820/SAR443820
Number analyzed (Participants) | 100 | 196
score on a scale
  Week 76 | 155.54 (92.17) | 144.91 (82.04)
  Week 104: number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Part B:Change From Baseline to Weeks 52, 76, and 104 in the Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) Total Score
Description: The ALSFRS-R is an instrument to evaluate the functional status of participants with ALS. It consists of 12 items across 4 sub-domains of bodily function: bulbar, fine motor, gross motor, and breathing. Each item was scored on an ordinal scale from 0 (total loss of function) to 4 (no loss of function). The total scores was the sum of the individual items score and it ranges from 0 to 48, with a higher score indicating better function. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) and Weeks 52, 76 and 104
Population: The ITT population consisted of all randomized participants. Only participants with data collected at specified timepoints are reported. The study was terminated prematurely since the Part A did not meet the primary endpoint. The data for Week 104 was not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 23 | 53
score on a scale
  Week 52 | -11.9 (7.8) | -12.1 (8.0)
  Week 76: number analyzed (Participants) | 3 | 7
  Week 76 | -12.0 (10.1) | -13.3 (9.0)
  Week 104: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Parts A and B: Change From Baseline to Weeks 24, 52, 76, and 104 in Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 Items (ALSAQ-5)
Description: The ALSAQ-5 is a patient-reported outcome that consists of 5 items derived from the ALSAQ-40. The 5 items closely resemble those of the 5-dimension scores of the ALSAQ-40: eating and drinking; communication; activities of daily living/independence; physical mobility; and emotional functioning. Each item was scored on a 5-point Likert scale ranging from 0 (never) to 4 (always or cannot do at all) according to the frequency of a particular problem. The total scores was the sum of the individual items score and it ranges from 0 to 20, with higher scores indicative of greater physical and emotional limitations. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) and Part A: Week 24, Part B: Weeks 52, 76 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 65 | 120 | 16 | 34
score on a scale
  Week 24: number analyzed (Participants) | 65 | 120 | 0 | 0
  Week 24 | 2.1 (3.1) | 2.4 (3.1) |  |
  Week 52: number analyzed (Participants) | 0 | 0 | 16 | 34
  Week 52 |  |  | 4.1 (4.2) | 4.4 (3.5)
  Week 76: number analyzed (Participants) | 0 | 0 | 3 | 4
  Week 76 |  |  | 5.0 (3.5) | 5.8 (5.3)
  Week 104: number analyzed (Participants) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: SAR443820; Analysis was performed using MMRM including treatment group, visit, randomization strata of the geographic region, ALS onset region, use of riluzole, use of edaravone, use of the combination of sodium phenylbutyrate and taurursodiol, treatment-by-visit interaction, disease duration, baseline ALSFRS-R score, baseline NfL, disease duration-by-visit interaction, and baseline ALSFRS-R score-by-visit interaction; Test type: Superiority; p = 0.2182, MMRM; LS Mean Difference = 0.520, 95% CI 2-sided [-0.310 to 1.350]

5. Secondary Outcome: Parts A and B: Change From Baseline to Weeks 24, 52, 76, and 104 in Percent Predicted Slow Vital Capacity (SVC)
Description: SVC is the maximum volume of air that can be slowly exhaled after slow, maximal inhalation. SVC is measured in participants while they are in an upright position at least 3 trials per assessment or up to 5 trials when the highest and second highest of the first 3 measurements differ by 10% or more. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) and Part A: Week 24, Part B: Weeks 52, 76 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of predicted volume
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 80 | 141 | 14 | 34
percentage of predicted volume
  Week 24: number analyzed (Participants) | 80 | 141 | 0 | 0
  Week 24 | -13.43 (14.66) | -11.24 (13.35) |  |
  Week 52: number analyzed (Participants) | 0 | 0 | 14 | 33
  Week 52 |  |  | -22.44 (16.35) | -18.29 (15.75)
  Week 76: number analyzed (Participants) | 0 | 0 | 3 | 5
  Week 76 |  |  | -31.30 (30.72) | -22.68 (15.93)
  Week 104: number analyzed (Participants) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: SAR443820; Analysis was performed using MMRM including treatment group, visit, randomization strata of the geographic region, ALS onset region, use of riluzole, use of edaravone, use of the combination of sodium phenylbutyrate and taurursodiol, treatment-by-visit interaction, disease duration, baseline SVC, baseline NfL, disease duration-by-visit interaction, baseline NfL-by-visit interaction, and baseline SVC-by-visit interaction; Test type: Superiority; p = 0.8134, MMRM; LS Mean Difference = 0.419, 95% CI 2-sided [-3.075 to 3.914]

6. Secondary Outcome: Parts A and B: Change From Baseline to Weeks 24 and 52 in Serum Neurofilament Light Chain (NfL)
Description: Serum blood samples were collected at indicated time points to measure changes in NfL, a marker of neuronal injury. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) and Part A: Week 24 and Part B: Week 52
Population: The ITT population consisted of all randomized participants. Only participants with data collected at specified timepoints are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 89 | 159 | 21 | 45
picograms per milliliter (pg/mL)
  Week 24: number analyzed (Participants) | 89 | 159 | 0 | 0
  Week 24 | 1.016 (5853.645) | 0.996 (6136.969) |  |
  Week 52: number analyzed (Participants) | 0 | 0 | 21 | 45
  Week 52 |  |  | 0.925 (-709.957) | 0.887 (-1488.592)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: SAR443820; Analysis was performed using MMRM including treatment group, visit, randomization strata of the geographic region, ALS onset region, use of riluzole, use of edaravone, use of the combination of sodium phenylbutyrate and taurursodiol, treatment-by-visit interaction, disease duration, log transformed baseline NfL, disease duration-by-visit interaction, and log transformed baseline NfL-by-visit interaction; Test type: Superiority; p = 0.2356, MMRM; Ratio of the LS Geometric Mean Ratios = 0.961, 95% CI 2-sided [0.899 to 1.027]

7. Secondary Outcome: Part A: Change From Baseline to Week 24 in Muscle Strength
Description: The muscles measured in the study included upper limb and lower-limb muscle groups. Bilateral hand grip were measured using a grip dynamometer and all other muscles were measured using a handheld dynamometer (HHD). Nine upper and lower extremity muscles or muscle groups were examined: shoulder flexion, elbow flexion, wrist extension, first dorsal interosseous contraction, hip flexion, knee extension, and ankle dorsiflexion. Each group was measured at least twice bilaterally and the average of the 2 highest measurements were analyzed. Individual muscles are standardized into the corresponding Z-scores using data from standard sample of healthy participants. A Z-score of 0 in a muscle measurement is equal to the mean of that measurement from the standard sample. Negative numbers indicate decreased muscle strength. For analysis, individual Z-scores were averaged to produce a total megascore including all available muscle groups. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) and Week 24
Population: The ITT population consisted of all randomized participants. Only participants with data collected at Baseline and Week 24 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 75 | 128
score on a scale | -0.498 (0.960) | -0.495 (0.704)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: SAR443820; Analysis was performed using MMRM including treatment group, visit, randomization strata of the geographic region, ALS onset region, use of riluzole, use of edaravone, use of the combination of sodium phenylbutyrate and taurursodiol, treatment-by-visit interaction, disease duration, baseline megascore, baseline NfL, disease duration-by-visit interaction, baseline NfL-by-visit interaction and baseline megascore-by-visit interaction; Test type: Superiority; p = 0.9565, MMRM; LS Mean difference = -0.005, 95% CI 2-sided [-0.193 to 0.183]

8. Secondary Outcome: Part B: Time From Baseline to Occurrence of Either Death or Permanent Assisted Ventilation
Description: The survival endpoint was defined as the time to death or permanent assisted ventilation (>22 hours a day for >7 consecutive days), whichever comes first. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) up to early termination of study, approximately 84 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 17 | 31
weeks | 31.90 (16.71) | 31.54 (18.82)

9. Secondary Outcome: Part B: Time From Baseline to the Occurrence of Death
Description: Time to the occurrence of death from baseline due to any reason has been reported. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) up to early termination of study, approximately 84 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 14 | 23
weeks | 38.30 (16.45) | 29.93 (17.13)

10. Secondary Outcome: Parts B and A+B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) After SAR443820 Initiation
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were defined as the AEs that developed, worsened or became serious during the treatment-emergent period (defined as time from first administration of study treatment (Day 1) to last administration of study treatment + 14 days). Serious adverse events (SAE): Any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. All TEAE occurring after SAR443820 initiation are provided for both randomized treatment arms in this endpoint.
Time Frame: From first dose of SAR443820 up to 14 days after last dose of SAR443820 administration in Part B, approximately 82 weeks for Parts A+B combined Arm (SAR443820/SAR443820), approximately 58 weeks for Part B Arm (Placebo/SAR443820)
Population: The safety population consisted of all randomized participants who received at least 1 dose (including partial dose) of SAR443820. All participants from safety population and treated with SAR443820 are included in Part B arm and participants from safety population are included in Parts A+B arm. The combined safety analysis for TEAE provided the accurate summary of all TEAE in both treatment groups after the initiation of SAR443820.
Measure: Count of Participants; unit: Participants
Groups:
- Part B (Placebo/SAR443820): Participants who had received placebo matching to SAR443820 tablet in Part A for 24 weeks, continued to receive first intake of SAR443820 20 mg tablet orally BID up to 80 weeks during Part B.
- Parts A+B: SAR443820/SAR443820: Participants who had received SAR443820 tablet in Part A for 24 weeks, continued to receive SAR443820 20 mg tablet orally BID up to 80 weeks during Part B.
Arm/Group | Part B (Placebo/SAR443820) | Parts A+B: SAR443820/SAR443820
Number analyzed (Participants) | 79 | 202
Participants
  TEAEs | 51 | 183
  TESAEs | 13 | 53

11. Secondary Outcome: Parts A and B: Plasma Concentration of SAR443820
Description: Plasma samples were collected at specified timepoints to determine plasma concentrations of SAR443820.
Time Frame: Part A: Day 1: 0.25- 1 hour and 1-3 hours post-dose; Weeks 2 and 8: pre-dose; Week 8: 0.25-3 hours post-dose; Part B: Week 28: pre-dose
Population: Pharmacokinetic (PK) population consisted of all randomized participants who received at least 1 dose of SAR443820 and had at least 1 PK assessment with adequate documentation of dosing and sampling. It was prespecified (statistical analysis plan) that participants will be analyzed according to actual intervention received. In Part B, all participants received SAR443820, so data were combined. Only participants who received SAR443820 with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram (ng)/mL
Units Other Than Participants: Samples
Groups:
- Part B: SAR443820: Participants received SAR443820 20 mg tablet orally BID for 80 weeks in Part B.
Arm/Group | Part A: SAR443820 | Part B: SAR443820
Number analyzed (Participants) | 202 | 252
Number analyzed (Samples) | 911 | 127
nanogram (ng)/mL
  Day 1: 0.25- 1 hours post-dose: number analyzed (Participants) | 202 | 0
  Day 1: 0.25- 1 hours post-dose: number analyzed (Samples) | 170 | 0
  Day 1: 0.25- 1 hours post-dose | 181.500 (169.940) |
  Day 1: 1-3 hours post-dose: number analyzed (Participants) | 202 | 0
  Day 1: 1-3 hours post-dose: number analyzed (Samples) | 199 | 0
  Day 1: 1-3 hours post-dose | 250.188 (95.867) |
  Week 2: pre-dose: number analyzed (Participants) | 202 | 0
  Week 2: pre-dose: number analyzed (Samples) | 186 | 0
  Week 2: pre-dose | 165.833 (91.355) |
  Week 8: pre-dose: number analyzed (Participants) | 202 | 0
  Week 8: pre-dose: number analyzed (Samples) | 177 | 0
  Week 8: pre-dose | 165.089 (92.686) |
  Week 8: 0.25- 3 hours post-dose: number analyzed (Participants) | 202 | 0
  Week 8: 0.25- 3 hours post-dose: number analyzed (Samples) | 179 | 0
  Week 8: 0.25- 3 hours post-dose | 365.488 (198.609) |
  Week 28: pre-dose: number analyzed (Participants) | 0 | 252
  Week 28: pre-dose: number analyzed (Samples) | 0 | 127
  Week 28: pre-dose |  | 171.865 (104.304)

12. Primary Outcome: Part A: Change From Baseline to Week 24 in the Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) Total Score
Description: The ALSFRS-R is an instrument to evaluate the functional status of participants with ALS. It consists of 12 items across 4 sub-domains of bodily function:
  bulbar, fine motor, gross motor, and breathing. Each item was scored on an ordinal scale from 0 (total loss of function) to 4 (no loss of function). The total scores was the sum of the individual items score and it ranges from 0 to 48, with a higher score indicating better function. The analysis was performed using mixed-effect model with repeated measures (MMRM). Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1, pre-dose) and Week 24
Population: The Intent-to-treat (ITT) population consisted of all randomized participants. Only participants with data collected at Baseline and Week 24 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 87 | 169
score on a scale | -5.9 (5.9) | -6.1 (5.4)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: SAR443820; Analysis was performed using MMRM including treatment group, visit, randomization strata of the geographic region, ALS onset region, use of riluzole, use of edaravone, use of the combination of sodium phenylbutyrate and taurursodiol, treatment-by-visit interaction, disease duration, baseline ALSFRS-R score, baseline serum neurofilament light chain (NfL), disease duration-by-visit interaction, baseline NfL-by-visit interaction and baseline ALSFRS-R score-by-visit interaction; Test type: Superiority; p = 0.5289, MMRM; Least Square (LS) Mean Difference = -0.414, 95% CI 2-sided [-1.706 to 0.878]

13. Primary Outcome: Part B: Combined Assessment of the Function and Survival (CAFS) Score at Week 52
Description: The CAFS at Week 52 is a composite endpoint based on time to earlier occurrence of death or permanent assisted ventilation (>22 hours a day for >7 consecutive days) and change from baseline in ALSFRS-R score up to Week 52. ALSFRS-R is a rating scale where 12 functions are rated on 5-point scales (from 0 to 4) with a maximum score of 48 (sum of all 12 items), with a higher score indicating better function. Each participant's outcome was compared to every other participant's outcome by time to death or permanent assisted ventilation and change on ALSFRS-R if survived without permanent assisted ventilation, assigned a score which is sum of comparisons (+1 [better], 0 [tie], -1 [worse]), and summed scores were ranked, from 1 to 296 (modified ITT[mITT] population) lowest rank corresponds to participant who died first and highest rank to 1 with best ALSFRS-R outcome among those who survived. A higher rank is considered a better outcome.
Time Frame: Week 52
Population: The mITT population consisted of all randomized participants who either died or had available baseline and at least 1 post-baseline ALSFRS-R assessment. All participants who had either early termination or who did not enter Part B, were also included in Week 52 analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo/SAR443820: Participants who had received placebo matching to SAR443820 tablet in Part A for 24 weeks, continued to receive SAR443820 20 mg tablet orally BID for 80 weeks during Part B.
  All death participants were automatically included in this analysis, irrespective whether they reached Week 52 or not.
- SAR443820/SAR443820: Participants who had received SAR443820 tablet in Part A for 24 weeks, continued to receive SAR443820 20 mg tablet orally BID for 80 weeks during Part B.
  All death participants were automatically included in this analysis, irrespective whether they reached Week 52 or not.
Arm/Group | Placebo/SAR443820 | SAR443820/SAR443820
Number analyzed (Participants) | 100 | 196
score on a scale | 154.89 (92.16) | 145.24 (82.09)
Statistical Analysis 1: Comparison: Placebo/SAR443820 vs SAR443820/SAR443820; Analysis was performed using rank analysis of covariance (ANCOVA) model including treatment group, randomization strata of the geographic region of the study site, ALS onset region (bulbar or other areas), use of riluzole (yes or no), use of edaravone (yes or no), use of the combination of sodium phenylbutyrate and taurursodiol (yes or no), disease duration (from first symptom onset to the screening visit), baseline ALSFRS-R score and baseline NfL; Test type: Superiority; p = 0.1830, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment (Day 1) up to 14 days after last dose of study treatment administration, up to 26 weeks for Part A, and 58 weeks for Part B. All-cause mortality (death) was assessed from signing of the informed consent form to study termination, approximately 99 weeks.
Description: Analysis was performed on safety population.
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
All-Cause Mortality (participants affected / at risk) | 5/102 | 11/202 | 9/79 | 12/136
Serious Adverse Events (participants affected / at risk) | 17/102 | 34/202 | 17/79 | 26/136
Other Adverse Events (participants affected / at risk) | 56/102 | 116/202 | 29/79 | 43/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=102) | Part A: SAR443820 (N=202) | Part B: Placebo/SAR443820 (N=79) | Part B: SAR443820/SAR443820 (N=136)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 2 (3)
Pneumonia Aspiration (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Skin Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suspected Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Speech Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left Ventricular Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 3 (3) | 12 (12)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T Wave Inversion (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 5 (5) | 3 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniofacial Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scapula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=102) | Part A: SAR443820 (N=202) | Part B: Placebo/SAR443820 (N=79) | Part B: SAR443820/SAR443820 (N=136)
Covid-19 (Infections and infestations) | 9 (9) | 20 (20) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (6) | 8 (8) | 5 (6) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 12 (13) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 25 (28) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (6) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10) | 14 (15) | 6 (6) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (10) | 13 (16) | 1 (1) | 8 (9)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (7) | 3 (3) | 3 (3)
Salivary Hypersecretion (Gastrointestinal disorders) | 6 (6) | 4 (4) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 11 (12) | 1 (1) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 2 (2) | 30 (32) | 10 (11) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 9 (13) | 11 (17) | 2 (5) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 22 (40) | 44 (91) | 10 (13) | 11 (12)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely since the Part A did not meet the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data

DOCUMENTS (2):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT05237284/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05237284/SAP_001.pdf